CLINICAL TRIAL: NCT05022030
Title: First-line Treatment of mCapOX Plus Cetuximab Versus mFOLFOX6 Plus Cetuximab for Metastatic Left-sided CRC Patients With Wild-type RAS/BRAF Genes: a Multicenter, Randomised, Phase 2 Study
Brief Title: First-line mCapOX+Cetuximab vs. mFOLFOX6+Cetuximab for Metastatic Left-sided CRC With Wild-type RAS/BRAF Genes
Acronym: CAPCET
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: West China Hospital (Other)
Collaborators: First Affiliated Hospital of Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Meng Qiu, Dr., West China Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20210602
Record Dates: First submitted 2021-08-23; First posted 2021-08-26 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-03

CONDITIONS: Colo-rectal Cancer; Capecitabine; Cetuximab
MeSH Terms: conditions — Colonic Neoplasms | interventions — Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental): mCapOX (capecitabine+oxaliplatin) plus cetuximab
  Interventions: Drug: mCapOX plus cetuximab
- Arm B (Active Comparator): mFOLFOX6 (fluorouracil+leucovorin+oxaliplatin) plus cetuximab
  Interventions: Drug: mFOLFOX6 plus cetuximab

INTERVENTIONS:
Drug: mCapOX plus cetuximab — capecitabine 1000mg/m2 po bid d1-7+oxaliplatin ivgtt 85mg/m2 d1+cetuximab ivgtt 500mg/m2, q2w
  Arms: Arm A
Drug: mFOLFOX6 plus cetuximab — oxaliplatin ivgtt 85mg/m2 d1+ leucovorin ivgtt 400mg/m2 d1+ fluorouracil iv bolus 400mg/m2 d1+ fluorouracil 2400mg/m2 continuous infusion for 46h+cetuximab ivgtt 500mg/m2, q2w
  Arms: Arm B

SUMMARY:
This prospective, randomized, phase 2 study is conducted to evaluate the efficacy and safety of first line mCapOX plus cetuximab versus mFOLFOX6 plus cetuximab for metastatic left-sided CRC patients with wild-type RAS and BRAF genes.

DETAILED DESCRIPTION:
The patients, who meet the inclusion criteria and have signed the informed consent, will be randomly assigned (1:1 ratio) to receive mCapOX plus cetuximab regimen (arm A) and mFOLFOX6 plus cetuximab regimen (arm B).

ELIGIBILITY:
Inclusion Criteria:

* Able to provide written informed consent and can understand and comply with the requirements of the study;
* Men and women ≥ 18 years of age;
* Patients with histologically or cytologically confirmed metastatic left-sided colorectal adenocarcinoma with wild-type RAS and BRAF genes;
* Presence of at least one evaluable lesion, as defined in RECIST Version 1.1;
* With an Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 1;
* No palliative first-line chemotherapy, targeted, immunotherapy, or prior platinum-based adjuvant chemotherapy, relapse more than 12 months from the end of adjuvant chemotherapy;
* According to the imaging findings and surgical assessment of initial unresectable, synchronous metastatic colorectal cancer, no serious complications of the primary tumor (obstruction, perforation, massive hemorrhage that cannot be treated in internal medicine, etc.) ;
* Life expectancy of longer than 3 months ( clinical assessment);
* Requirements for lab indicators neutrophils ≥ 1.5 × 109/L, platelets ≥ 75 × 109/L, hemoglobin ≥ 8 g/dL, total bilirubin ≤ 1.5 × upper limit of normal (UNL); ASAT (SGOT) and/or ALAT (SGPT) ≤ 2.5 × UNL (≤ 5 × UNL if liver metastases); alkaline phosphatase ≤ 2.5 × UNL (≤ 5 × UNL if liver metastases, ≤ 10 × UNL if bone metastases); LDH < 1500 U/L; creatinine clearance (calculated according to Cockcroft and Gault formula) > 50 mL/min or serum creatinine ≤ 1.5 × UNL;

Exclusion Criteria:

* Patients with mCRC who were initially resectable with R0 resection or radiofrequency or SBRT were excluded.
* Patients diagnosed with MSI-H or dMMR by PCR or immunohistochemistry
* Hypersensitivity to any therapeutic agent.
* Patients who received adjuvant chemotherapy containing oxaliplatin and fluorouracil within 12 months before entering the study;
* Patients who have failed one or more palliative chemotherapy regimens;
* Patients with uncontrolled hepatitis B virus
* Peripheral neuropathy ≥ CTC grade 2;
* Neurological or psychiatric disorders affecting cognitive performance;
* Patients with central nervous system metastasis could not be controlled with radiotherapy;
* Previous enteritis, chronic diarrhea, or recurrent bowel obstruction; uncontrolled bleeding from internal medicine; bowel perforation
* Uncontrolled concomitant diseases within 6 months before the study, including unstable angina, acute myocardial infarction, cerebrovascular accident, etc.;
* Pregnant or lactating patients, or those of childbearing potential who do not take adequate contraceptive measures;
* History of other malignancies, but no disease-free survival longer than 5 years;
* Patients concurrently receiving other anti-tumor treatment or participating in other interventional clinical trials;
* Patients who are unable to comply with this study for psychological, family or social reasons.
* Patients with other serious diseases that the investigator considers not suitable.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2021-07-21 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) rate at 9 months | 9 months
  PFS rate at 9 months is defined as the proportion of patients without PD or death at 9 months after randomization.

SECONDARY OUTCOMES:
Objective response rate | 6 months
  The rate of complete response and partial response
Disease control rate | 6 months
  The rate of complete response, partial response and stable disease.
Progression free survival | up to 3 years
  Progression free survival is defined as the period from randomization to disease progress or death.
Overall survival | up to 4 years
  Overall survial is defined as the period from randomization to death.
Adverse event rate | 3 years
  The rate of adverse event after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Meng Qiu, M.D., Principal Investigator — West China Hospital
Locations (1):
- West China Hospital of Sichuan University, Chengdu, Sichuan, China